CLINICAL TRIAL: NCT05749029
Title: An Online, Compassion Intervention to Improve Shame, Self-criticism, and Physical Wellbeing in Adults with Type 1 and Type 2 Diabetes Mellitus (T1DM; T2DM)
Brief Title: An Online, Compassion Intervention for Adults with Type 1 and Type 2 Diabetes Mellitus (T1DM; T2DM).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Principal Investigator, Hetashi Bawa, Trainee Clinical Psychologist, Canterbury Christ Church University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hetashi Bawa MRP 2021
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Compassion Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All the outcome measures will be self-report questionnaires that will be completed by an online automated system with no involvement of the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Four Week Self-Compassion Course
- Waitlist Control (No Intervention): Control participants will receive no intervention during the study but will be given the option of accessing the online self-compassion intervention after the study is complete.

INTERVENTIONS:
Behavioral: Four Week Self-Compassion Course — This is a four-week self-compassion course supplied by Balanced Minds. The owner of Balanced Minds is a Consultant to this study, who will be providing access to participants.
  The self-help, self-compassion course is based on Compassionate Mind Training. This provides participants with opportunities to develop skills and attributes of compassion through a weekly 30-minute video on a specified topic, a 10-minute compassionate exercise that participants are encouraged to engage in daily for the week and a brief summary of the compassionate topic. The topics of the course are:
  1. The Foundations of Self-Compassion
  2. Developing your Compassionate Self
  3. Deepening the Compassionate Relationship with Yourself
  4. Self-compassion in Everyday Life.
  Other Names: Online Self-Compassion Course
  Arms: Intervention

SUMMARY:
The goal of this research study is to evaluate a programme that is based on Compassionate Mind Training (CMT) over four-weeks. The programme intends to share information and strategies to reduce diabetes distress, self-criticism, and shame, and improve physical health in people who have Type 1 and Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
This Randomised Controlled Trial (RCT) will compare a CMT intervention for people with Type 1 and Type 2 Diabetes Mellitus with a waitlist control group who will be given access after the study.

The outcome measures will be completed at baseline (week 0), post-intervention (week 4), and at follow-up (week 8).

ELIGIBILITY:
Inclusion Criteria:

* Resident in the United Kingdom;
* Clinician diagnosed Type 1 Diabetes Mellitus or Type 2 Diabetes Mellitus;
* Self-managing condition;
* Diabetes diagnosed over a year ago.

Exclusion Criteria:

* Diagnosis of Gestational Diabetes or Pre-Diabetes.
* Current severe mental health condition;
* Currently self-harming or suicidal;
* Currently engaging in psychological therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes Distress Scale (DDS) scores from baseline (week 0) to post-intervention (week 4). | Post-intervention (week 4)
  The DDS is a 17-item measure of problems and hassles related to diabetes.
  The DDS establishes a total mean score and a mean score for its four sub-scales. Scores will range from 1 to 6. Mean scores of 3 or above is considered distress worthy of clinical attention.

SECONDARY OUTCOMES:
Change in the total score on the External and Internal Shame Scale (EISS) from baseline (week 0) to post-intervention (week 4). | Post-intervention (week 4)
  The EISS is an eight-item scale measuring external and internal dimensions of shame.
  Higher scores indicate higher levels of shame and a total score varies between 8 and 40.
Change in Forms of Self-Criticising/Attacking and Self-Reassuring Scale (FSCRS) scores from baseline (week 0) to post-intervention (week 4). | Post-intervention (week 4)
  The FSCRS is a 22-item scale with statements measuring inadequate self, hated self and reassured self.
  Scores will range from 0 to 88.
Change in Fears of Compassion Scale (FCS) scores from baseline (week 0) to post-intervention (week 4). | Post-intervention (week 4)
  The FCS is a 15-item measure of fear of compassion towards self.
  Scores will range from 0 to 60. Higher scores indicate greater fear of compassion.
Change in Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS) scores at baseline (week 0) and post-intervention (week 4). | Post-intervention (week 4)
  14-item measure assessing mental wellbeing in the non-clinical sample. Scores on the WEMWBS will range from 14 to 70. Higher scores indicate greater positive mental wellbeing.
Change in Compassionate Engagement and Action Scale (CEAS) scores at baseline (week 0) and post-intervention (week 4). | Post-intervention (week 4)
  The CEAS is a 13-item measure of compassionate engagement and action.
  The engagement sub-scale will establish a score between 6 and 60.
  The action sub-scale will establish a score between 4 and 40.
Change in HbA1c from baseline (week 0) to follow-up (week 8). | Follow-up (week 8)
  Participants will be asked to self-report a blood glucose (HbA1c) level taken by a healthcare provider in the past three to six months at baseline and at one-month post-intervention.
  Higher HbA1c levels indicate poorer diabetes control.
Change in Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS) scores at baseline (week 0) and follow-up (week 8). | Follow-up (week 8)
  Please see description above.
Change in the total score on the External and Internal Shame Scale (EISS) from baseline (week 0) to follow-up (week 8). | Follow-up (week 8)
  Please see description above.
Change in Forms of Self-Criticising/Attacking and Self-Reassuring Scale (FSCRS) scores from baseline (week 0) to follow-up (week 8). | Follow-up (week 8)
  Please see description above.
Change in Diabetes Distress Scale (DDS) scores from baseline (week 0) to follow-up (week 8). | Follow-up (week 8)
  Please see description above.
Change in Fears of Compassion Scale (FCS) scores from baseline (week 0) to follow-up (week 8) | Follow-up (week 8)
  Please see description above.
Change in Compassionate Engagement and Action Scale (CEAS) scores at baseline (week 0) to follow-up (week 8). | Follow-up (week 8)
  Please see description above.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Hebben-Wadey, DClinPsy, Study Director — Canterbury Christ Church University; Hetashi Bawa, BSc, MSc, Principal Investigator — Canterbury Christ Church University
Locations (1):
- Salomons Institute for Applied Psychology, Canterbury Christ Church University, 1 Meadow Road, Royal Tunbridge Wells, Tunbridge Wells, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data would be made available to researchers on reasonable request after the study findings have been published.